CLINICAL TRIAL: NCT01550419
Title: Effect of Atorvastatin on the Frequency of Ventilator-associated Pneumonia in Patients With Ischemic Stroke
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Minhang Central Hospital (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Liu Chunyan, Department of Intensive Care Unit, Minhang Central Hospital, Shanghai Minhang Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MHC Hospital 01
Record Dates: First submitted 2012-03-02; First posted 2012-03-12 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Ventilator-associated Pneumonia; Ischemic Stroke
Keywords: Ventilator-associated pneumonia; Ischemic stroke; Atorvastatin; Morbidity; Mortality
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Ischemic Stroke | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin(50 characters) (Experimental)
  Interventions: Drug: Atorvastatin
- Placebo(50 characters) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Patients will receive 40mg atorvastatin(one tablet) over night via enteral feeding tube or per os during they stay in ICU at most thirty days.
  Other Names: Lipitor
  Arms: Atorvastatin(50 characters)
Drug: Placebo — The smell and shape of placebo are the same as atorvastatin
  Other Names: No other name
  Arms: Placebo(50 characters)

SUMMARY:
Ventilator-associated pneumonia (VAP) is an important cause of morbidity and mortality in ventilated critically ill patients specially in intensive care unit (ICU). It is associated with an increased duration of mechanical ventilation, high death rates and increased healthcare costs in China. However, VAP is preventable and many practices have been demonstrated to reduce the incidence of this disease, but the morbidity is still so high. So much more methods of prevention should be needed to reduce the incidence of VAP.

Statins (3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitors) present anti-inflammatory and immunomodulatory effects besides their ability to regulate cholesterol composition. So it is hypothesized that early use of statin may prevent some of the infection disease such as VAP.

Actually, Two studies have showed that statin treatment is associated with reduced risk of pneumonia. However, the relationship between statins and reduced risk of pneumonia is not consistent.

After reviewing some of the guidelines,meta analyses and system reviews, the investigator find that advanced age,immune suppression from disease or medication and specially depressed level of consciousness are the risk factors of VAP. So the investigator assumes that early use of statin may give us a favorable outcome in the patients with coma or in the patients with severe disease (Acute Physiology and Chronic Health Evaluation II score > 15 or Glasgow coma score < 7).

In addition there is no prospective study to investigate the role of statins in VAP in the patients with ischemic stroke. The investigator hopes that this study can approve the relationship between statins and reduced risk of VAP in the patients with ischemic stroke. And it can improve the processes,outcomes and costs of critical care as well.

DETAILED DESCRIPTION:
This is a one-center, two-arm, randomized, single-blinded, controlled trial. When a patient with ischemic stroke who needs mechanic ventilation is admitted to ICU,a sealed envelop will be opened which decide whether the patient is assigned to the placebo arm or the atorvastatin arm. During they stay in ICU, one tablet of atorvastatin (40mg) or one tablet of placebo will be administered. Atorvastatin or placebo will be administered through an enteral feeding tube or administered orally when patients are able to safely take oral medications.

VAP diagnosis accords with the comprehensive evidence-based clinical practice guidelines for ventilator-associated pneumonia:Diagnosis and treatment which was published in 2008.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with ischemic stroke who are admitted to Intensive Care Unit(ICU) between 1st March.2012 at 00:00 hours (midnight) and the finish date of 31st March. 2014 at 23:59 hours (11.59 pm). Patients who are already in the ICU prior to 1st March. 2012 at 00:00 hours will not be included in the study.
* Duration of mechanical ventilation > 48h through tracheal tube or tracheotomy
* Informed consent

Exclusion Criteria:

* Patients with pneumonia when they are admitted to ICU.
* Previous use of statin for cholesterol regulation.
* Chronic liver disease or active liver disease.
* Increase of CPK (over 3 times the upper limit) during hospitalization.
* Malnutrition.
* Pregnancy.
* Unwilling to continue the therapy during hospitalization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative frequency of ventilator-associated pneumonia | 30 days

SECONDARY OUTCOMES:
Mortality | 30 days
Ventilation free days | 30 days
Antibiotic free days | 30 days
Whether the bacteria of multidrug-resistance can be isolated from the sputum culture | 30 days
  We will find whether methicillin-resistant Staphylococcus aureus(MRSA), extended-spectrum beta-lactamase(ESBLs) or Vancomycin-resistant enterococcus (VRE)can be isolated from the sputum culture.
Adverse effects | 30 days
  Creatine kinase of more than three times the upper normal limit or hepatic enzyme dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Liu ChunYan, MD, Principal Investigator — Shanghai Minhang Central Hospital
Locations (1):
- Shanghai Minhang Central Hospital, Shanghai, China